CLINICAL TRIAL: NCT00425997
Title: A 10-week Multicenter,Forced-titration Study Using 24-hr ABPM to Evaluate the Efficacy of Valsartan/Hydrochlorothiazide (HCTZ) Treatment Regimen vs Conventional Treatment Regimen With Amlodipine and Hydrochlorothiazide (HCTZ) in Patients With Stage 2 Hypertension
Brief Title: Efficacy of Valsartan/Hydrochlorothiazide Versus Amlodipine and Hydrochlorothiazide in Patients Hypertension
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Study director, Novartis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CVAH631BUS07
Record Dates: First submitted 2007-01-23; First posted 2007-01-24 (Estimated); Last update posted 2011-06-08 (Estimated); Status verified 2011-06

CONDITIONS: Hypertension
Keywords: Hypertension, valsartan/HCTZ, amlodipine and HCTZ
MeSH Terms: conditions — Hypertension | interventions — Amlodipine; Hydrochlorothiazide

INTERVENTIONS:
Drug: Valsartan/HCTZ
Drug: amlodipine
Drug: HCTZ

SUMMARY:
This study will evaluate the efficacy of valsartan/hydrochlorothiazide versus amlodipine and hydrochlorothiazide in patients with Stage 2 hypertension using 24-hr ambulatory blood pressure monitoring (ABPM)

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients 18 years of age or older
* Diagnosed of having hypertension, defined as a mean seated systolic BP ≥160 mmHg (Stage 2 hypertension)

Exclusion Criteria:

* Symptomatic or severe hypertension
* Patients treated with more than 2 antihypertensive medications
* Clinically known or suspected history of secondary hypertension
* Myocardial infarction, stroke, transient ischemic attack, cardiovascular revascularization/angioplasty in last 6 months
* Diagnosis of heart failure (NYHA Class II-IV)
* Chronic renal or severe hepatic disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 480 (Estimated)
Dates: Start 2006-12; Primary Completion 2007-10 (Actual); Study Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
-Change from baseline in mean 24-hr ambulatory systolic blood pressure (BP) after 10 weeks of treatment of valsartan/HCTZ versus amlodipine and HCTZ

SECONDARY OUTCOMES:
change from baseline in mean 24-hr ambulatory diastolic BP and pulse pressure after 10 weeks of treatment of valsartan/HCTZ versus amlodipine and HCTZ
Change from baseline in mean seated systolic and diastolic BP after 10 weeks of treatment of valsartan/HCTZ versus amlodipine and HCTZ
Compare the proportion of patients achieving blood pressure goal and tolerability after 10 weeks of treatment of valsartan/HCTZ versus amlodipine and HCTZ

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Chair — Sponsor GmbH
Locations (1):
- Sites in USA, East Hanover, New Jersey, United States

REFERENCES:
- [Derived] Raij L, Egan BM, Zappe DH, Purkayastha D, Samuel R, Sowers JR. Office and ambulatory blood pressure-lowering effects of combination valsartan/hydrochlorothiazide vs. hydrochlorothiazide-based therapy in obese, hypertensive patients. J Clin Hypertens (Greenwich). 2011 Oct;13(10):731-8. doi: 10.1111/j.1751-7176.2011.00499.x. Epub 2011 Jul 14. PMID 21974760